CLINICAL TRIAL: NCT07126015
Title: Predicting Biological Therapy Effectiveness in Ulcerative Colitis Patients Using Intestinal Ultrasound and Visceral Fat Assessment: A Prospective Study
Brief Title: Predicting Biologic Therapy Success in Ulcerative Colitis Using Intestinal Ultrasound and Fat Assessment
Acronym: IBD/VAT
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Mohammed Abdel Mowgod, Lecturer of Tropical Medicine and Gastroenterology, Assiut University
Other Study IDs: 4-2025-300643
Record Dates: First submitted 2025-08-03; First posted 2025-08-15 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-08

CONDITIONS: Predicting Biologics Success Via VAT Assessment

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Our study aimed to detecting biological therapy effectiveness in UC patients using visceral fat assessment

DETAILED DESCRIPTION:
Ulcerative colitis (UC) has a relapsing-remitting course which necessitates frequent follow-up examinations to monitor disease activity.

Disease management was previously guided by patient reported symptoms, and treatment targets were based on symptom control. However, the patient's symptoms do not necessarily correspond to inflammatory activity and current guidelines recommend that management should be based on objective evaluations.

Gastrointestinal ultrasound [GIUS] has high diagnostic accuracy for detecting active CD, and in trained hands, it can make significant impact on clinical decision-making.

Furthermore, as it is non-invasive, readily available and can be performed bedside, the modality seems well suited for bedside and frequent activity monitoring.

UC is often associated with underweight (BMI < 18 kg/m2); however, numerous studies find overweight and obesity also common.

Patients were characterized by increased fat deposition and reduced skeletal muscles and theses patients are refractory to IBD treatment may have an increased risk of sarcopenic obesity.

Visceral adipose tissue (VAT) is the white adipose tissue surrounding the viscera, which can be divided into omental adipose tissue, mesenteric adipose tissue (MAT), retroperitoneal fat, peri-gonadal fat, and pericardial fat.

VAT releases inflammatory mediators, such as TNF-α, which are closely associated with inflammation. This suggests that VAT plays an inflammatory role in UC pathogenesis; arguably, VAT is one of the radiological markers.

One research found that VAT is associated with mucosal healing of anti-TNF therapy in Crohn's disease (CD). Studies demonstrated that a higher ratio of visceral to subcutaneous fat (SAT) (VAT:SAT) is linked to a shorter time to IBD flare-ups, including in ulcerative colitis.

Some research indicates that higher VAT levels might be associated with poorer responses to certain IBD treatments, potentially due to the inflammatory environment created by visceral fat.

ELIGIBILITY:
Inclusion Criteria:

* Any patient above age of 18 years old and diagnosed to have active UC through
* Clinical features: rectal bleeding, with frequent stools and mucous discharge from the rectum. Some patients also describe tenesmus. The onset is typically insidious.
* Endoscopic findings include the following; loss of vascular pattern, Granular and fragile mucosa, friability, ulcerations, erosions, pseudo-polyposis.

Exclusion Criteria:

* Patients with UC who are under age of 18 years old.
* Pregnancy.
* Previous colectomy.
* Patient refuse to participate in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with ulcerative colitis will undergo detailed medical history (abdominal pain, bloody diarrhea frequency, tenesmus, mucus in stool), anthropometric measurements (weight, height, waist circumference, BMI), and physical examination for fever, tachycardia, abdominal tenderness, and weight loss. Disease activity will be assessed using Montreal classification, Harvey Bradshaw Index (HBI < 5 = remission), and Truelove & Witts criteria. Visceral adipose tissue volume and distribution will be evaluated by abdominal and pelvic CT examination.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Visceral Adipose Tissue Volume Measured by abdominal and pelvic CT examination from Baseline to month 6 | Baseline (pre-treatment) and after induction dose (typically 6 month post-initiation of biological therapy) by abdominal and pelvic CT examination
Effectiveness of Biological Therapy in UC Patients Based on Changes in Visceral Adipose Tissue (VAT) by abdominal and pelvic CT examination | Baseline (pre-treatment) and after induction dose (typically 6 month post-initiation of biological therapy)
  Change in visceral fat volume and distribution as assessed by abdominal and pelvic CT examination before and after the induction phase of biological therapy in patients with ulcerative colitis. CT scans will be analyzed to determine the relationship between VAT and treatment response, considering clinical and endoscopic outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Amira M Abdelmawgod, Lecturer, Tropical Medicine, Principal Investigator — Assiut University